CLINICAL TRIAL: NCT00181753
Title: Study of Glutamate and Glutamine Metabolism in Burn Patients Receiving Enteral or Parenteral Nutrition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: State of Mass. tightened regulations for making intravenous solutions for research subjects. Study was withdrawn and no participants were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ronald G. Tompkins, MD, ScD, Chief, Burn Service, Massachusetts General Hospital
Organization: National Institute of General Medical Sciences (NIGMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2P50GM021700-27A1 (NIH); 2004-P-001946
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Burns
Keywords: glutamine metabolic kinetics; glutamate metabolic kinetics; enteral nutrition; parenteral nutrition; burn injury; stable isotopes
MeSH Terms: conditions — Burns; Hyperphagia | interventions — Parenteral Nutrition; Nutritional Support; Glutamine; Glutamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Burn Patients receiving at least 3 days of parenteral feeding on routine formula
  Interventions: Drug: standard vs. glutamine enteral or parenteral feeding.; Dietary Supplement: Stable isotope tracer study; Dietary Supplement: Stable isotope study
- 2 (Experimental): Burn patients receiving at least 3 days on parenteral feeding on glutamine enriched formula.
  Interventions: Drug: standard vs. glutamine enteral or parenteral feeding.; Dietary Supplement: Stable isotope tracer study; Dietary Supplement: Stable isotope study
- 3 (Experimental): Burn patients receiving at least 3 days of enteral feeding on routine formula.
  Interventions: Drug: standard vs. glutamine enteral or parenteral feeding.; Dietary Supplement: Stable isotope tracer study; Dietary Supplement: Stable isotope study
- 4 (Experimental): Burn patients receiving at least 3 days of enteral feeding on glutamine-enriched formula.
  Interventions: Drug: standard vs. glutamine enteral or parenteral feeding.; Dietary Supplement: Stable isotope tracer study; Dietary Supplement: Stable isotope study

INTERVENTIONS:
Drug: standard vs. glutamine enteral or parenteral feeding. — Patient in each group will continue on the same diet for > 3 days before we conduct stable isotope tracer measurements.
  Other Names: Nutritional Support; Glutamine; Glutamate; Amino Acide
Dietary Supplement: Stable isotope tracer study — 7 hours of primed constant infusion
  Other Names: Glutamine; Stable isotope study
Dietary Supplement: Stable isotope study — 7 hours of primed constant infusion of stable isotope tracers.
  Other Names: Stable isotopes; Glutamine
Dietary Supplement: Stable isotope tracer study — 7 hours of primed constant stable isotope tracer infusion.
  Other Names: Stable isotope tracers; Glutamine
Dietary Supplement: Stable isotope tracer study — 7 hours primed constant infusion of stable isotope tracer study
  Other Names: Glutamine; Stable isotope tracers

SUMMARY:
The purpose of the study is to understand how the body uses amino acids in burned patients during the time they cannot eat normally. Amino acids occur naturally in the body and the food we eat. The body combines amino acids to make protein. It uses the proteins to do things such as heal wounds, fight infection, and provide energy. We are studying two ways of receiving nutrition: through a vein or through a tube. We are also studying two different types of food: with or without glutamine. The results of this study will be used to determine the best type and way to supply nutrients during a severe burn injury. We hope to learn how to help the body use nutrients more efficiently to better repair wounded tissues and recover earlier from injury.

DETAILED DESCRIPTION:
We hypothesize that:

1. Burn patients will experience an increased conversion of glutamine to glutamate and a decreased conversion of glutamate to glutamine as compared to healthy subjects. The net direction is from glutamine to glutamate in burn patients and would render glutamine as a conditionally essential amino acid.
2. Because of the limited ability of liver to oxidize glutamate, it is possible that large doses of glutamine may cause increased gluconeogenesis in burn patients, thus aggravating the glucose homeostasis secondary to insulin resistance.
3. Enterally and parenterally fed glutamine and glutamate have different metabolic fate in the splanchnic bed and peripheral regions, therefore the doses should be tailored according to the route of administration.

This study, using stable isotope tracers, aims to track the metabolic fate of glutamine and glutamate in body with the goal of enhancing nutritional efficiency.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following:

  * 5% Total Body Surface Area Thermal Burn
* Inhalation Injury
* Resting Energy Expenditure of >15% of the predicted Basal Metabolic Rate Using Harris-Benedict.
* Receiving Enteral or Parental Nutritional Support

Exclusion Criteria:

* Pre-existing:
* Thyroid disease
* Congestive Heart Failure (Ejection fraction <20%)
* Malignancy currently under treatment
* Medical conditions requiring glucocorticoid treatment
* Decision not to treat because of severity of injury
* Presence of Anoxic brain injury with no expectation for recovery
* Self-Inflicted thermal injury
* Ileus, gut paralysis, or facial injuries
* No NG or OG tube as part of their clinical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
This is a nutritional study. The primary outcome is to measure the protein kinetics for metabolism of the amino acid, glutamate and glutamine. Fate will be determine from measurements of subject blood and air samples. | 3 days and above

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Tompkins, MD, ScD, Principal Investigator — MGH, Shriners Burn Hospital-Boston
Locations (1):
- Massachusetts General Hospital Burn Unit, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sheridan RL, Prelack K, Yu YM, Lydon M, Petras L, Young VR, Tompkins RG. Short-term enteral glutamine does not enhance protein accretion in burned children: a stable isotope study. Surgery. 2004 Jun;135(6):671-8. doi: 10.1016/j.surg.2003.11.014. PMID 15179374
- [Background] Young VR, Ajami AM. Glutamine: the emperor or his clothes? J Nutr. 2001 Sep;131(9 Suppl):2449S-59S; discussion 2486S-7S. doi: 10.1093/jn/131.9.2449S. PMID 11533293
- [Background] Herndon DN, Tompkins RG. Support of the metabolic response to burn injury. Lancet. 2004 Jun 5;363(9424):1895-902. doi: 10.1016/S0140-6736(04)16360-5. PMID 15183630